CLINICAL TRIAL: NCT04164927
Title: The Effects of Manual Lymphatic Drainage and Kinesiotaping on Lower Extremity Edema and Functional Outcomes in Patients With Total Knee Arthroplasty
Brief Title: The Effects of Manual Lymphatic Drainage and Kinesiotaping on Lower Extremity Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HANDE GUNEY, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO15-152
Record Dates: First submitted 2018-06-14; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Total Knee Arthroplasty; Edema; Exercise
MeSH Terms: conditions — Edema; Motor Activity | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Taping (Active Comparator): Lymphatic correction method is applied via Kinesiotaping depending on the size of the leg two or three fan-cut tape was applied with light paper-off tension on the frontal, medial and lateral aspects of the limb. Certified Kinesio Tape practitioner applied Kinesiotaping on the second day (day 2) post-surgery and once a week.
  Interventions: Other: Manual Lymphatic Drainage; Other: Control
- Manual Lymphatic Drainage (Active Comparator): A standardized 30-minute manual lymphatic drainage (MLD) treatment is applied to MLD group. On the second day (day 2) post-surgery, patients allocated to the MLD group underwent a standardized 30 minute MLD treatment on the operated limb by an experienced remedial massage therapist trained in delivering MLD.
  Interventions: Other: Kinesio Taping; Other: Control
- Control (No Intervention): Standard postoperative rehabilitation program is applied to Control Group. Knee-based exercises were undertaken in supine (active- assisted knee flexion using a bandage, inner range quadriceps contractions, and straight-leg raises), seated (active-assisted knee flexion using the contralateral limb and inner range quadriceps contractions), and standing (hip and knee flexion, active hamstring curls, lunges on a step, hamstring stretches) postures.

INTERVENTIONS:
Other: Manual Lymphatic Drainage — 1. Lymphatic correction method was used via the KinesioTaping® to patients group.
  2. Standardized 30-minute Manuel Lymphatic Drainage treatment was applied to the MLD group.
  3. Control group received only physiotherapy treatment.
  Arms: Kinesio Taping
Other: Kinesio Taping — Depending on the size of the leg two or three fan cut tapes were applied with light paper-off tension on the frontal, medial and lateral aspects of the limb. Kinesio taping was applied by certified Kinesio Tape practitioner once a week to Kinesiotaping group.
  Arms: Manual Lymphatic Drainage
Other: Control — Knee-based exercises were undertaken in supine (active- assisted knee flexion using a bandage, inner range quadriceps contractions, and straight-leg raises), seated (active-assisted knee flexion using the contralateral limb and inner range quadriceps contractions), and standing (hip and knee flexion, active hamstring curls, lunges on a step, hamstring stretches) postures. These exercises were undertaken in sets of 10 repetitions, 3 times daily; the physiotherapist was present to assist, as required, on 2 occasions per day for the first 3 postoperative days and then once daily from day 4 until hospital discharge.
  Arms: Kinesio Taping; Manual Lymphatic Drainage

SUMMARY:
Significant trauma and muscular tightness often result during Total Knee Arthroplasty (TKA) surgery and thus act to restrict tissue fluid movement resulting with lower extremity edema. Kinesio Taping® is applied directly on the skin for restoration of normal fluid perfusion, removing congestion of lymphatic fluid or hemorrhages. In addition Manual Lymphatic Drainage (MLD) enhances blood circulation and stimulates the lymphatic movement and unblocks lymphatic territories. The aim of the study was to investigate the effectiveness of Kinesio Taping® and MLD in reducing postoperative edema and pain in the early stage after TKA.

DETAILED DESCRIPTION:
Procedures: Patients who underwent unilateral TKA were randomized as Kinesio Taping® group, MLD group and control group. For all patients, postoperative rehabilitation program included early mobilization and physical therapy twice a day during the stay in orthopedic traumatology department. On the second day after surgery, lymphatic correction method was used on the Kinesio Taping® group patients and a standardized 30-minute MLD treatment was applied to the MLD group patients. Control group received only physiotherapy treatment. Circumference measurements were applied on preoperatively and the second, third, fourth day and 6th weeks after surgery. Knee Injury and Osteoarthritis Outcome Score (KOOS) was used to determine the functional outcomes on the 6th weeks after surgery. Repeated measures of variance analysis was used to determine time differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* TKA surgery

Exclusion Criteria:

* active infection
* malignant tumor
* major cardiac pathology, or thrombus or venous obstruction that was pre-diagnosed or revealed on a routine preadmission hospital screening

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Circumference measurements | This outcome measure is assessing a change from the postoperative day 2 at 3rd month after surgery
  Circumference measurements

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | This outcome measure is assessing a change from the postoperative day 2 at 3rd month after surgery
  Knee Injury and Osteoarthritis Outcome Score (KOOS) evaluates the functional status of knee joint. total points range between 0-100 points. higher points represents a better outcome. total score is the averaged subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Güney Deniz, assoc. prof., Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pichonnaz C, Bassin JP, Lecureux E, Christe G, Currat D, Aminian K, Jolles BM. Effect of Manual Lymphatic Drainage After Total Knee Arthroplasty: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 May;97(5):674-82. doi: 10.1016/j.apmr.2016.01.006. Epub 2016 Jan 30. PMID 26829760
- [Background] Ebert JR, Joss B, Jardine B, Wood DJ. Randomized trial investigating the efficacy of manual lymphatic drainage to improve early outcome after total knee arthroplasty. Arch Phys Med Rehabil. 2013 Nov;94(11):2103-11. doi: 10.1016/j.apmr.2013.06.009. Epub 2013 Jun 26. PMID 23810354